CLINICAL TRIAL: NCT07318519
Title: Cognitive Behavioral Theory-assisted Virtual Reality for Chronic Cancer Pain (VR-CAN): Device Prototype Development and Feasibility Testing
Brief Title: Cognitive Behavioral Theory-assisted Virtual Reality for Chronic CANcer Pain (VR-CAN)
Acronym: VR-CAN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medstar Health Research Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Device Feasibility
Other Study IDs: 1R21CA299799-01 (NIH); 1R21CA299799-01 (NIH)
Record Dates: First submitted 2025-06-25; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Cancer; Cancer Pain; Chronic Cancer Pain
Keywords: cancer; pain; chronic pain; cognitive behavioral therapy; virtual reality
MeSH Terms: conditions — Neoplasms; Cancer Pain; Pain; Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual reality delivered behavioral skills for pain management (Experimental): Participants use VR-CAN therapy at home, 10 minutes per session, daily for 14 days
  Interventions: Device: VR-CAN prototype chronic cancer pain therapy -- virtual reality program delivering CBT for chronic cancer pain management
- Tablet-based delivery of behavioral skills for pain management (Active Comparator): Participants use a two-dimensional skills-based intervention delivered by handheld tablet at home, 10 minutes per session, daily for 14 days
  Interventions: Device: Active Control -- two-dimensional tablet-delivered intervention

INTERVENTIONS:
Device: VR-CAN prototype chronic cancer pain therapy -- virtual reality program delivering CBT for chronic cancer pain management — VR-CAN participants will be instructed to use the prototype VR-CAN software on the VR device at home daily for two weeks, at least 10 minutes per session, beginning the day after enrollment.
  Arms: Virtual reality delivered behavioral skills for pain management
Device: Active Control -- two-dimensional tablet-delivered intervention — Tablet-based active control participants will follow the same prescription as the experimental arm (i.e., using assigned technology >10 min/daily for two weeks at home), except they will view a two-dimensional, non-CBT skills version using a tablet device.
  Other Names: Handheld tablet delivered two-dimensional skills based intervention
  Arms: Tablet-based delivery of behavioral skills for pain management

SUMMARY:
While chronic cancer pain affecting as many as 75% of patients is typically addressed using pharmacologic interventions, experts and patients alike support maximizing any relevant non-pharmacologic interventions as well, such as cognitive behavioral therapy. Virtual reality, a novel technology that can temporarily immerse users in a calm, pleasant environment, has been increasingly shown to facilitate improvement in different acute and chronic pain syndromes by providing distraction from pain and lowering pain sensation. To address the significant needs of patients living with chronic cancer pain, we aim to develop and pilot test a prototype device that will leverage cognitive behavioral therapy principles to deliver a novel virtual reality pain therapy. The investigators will do this through the following steps:

Step 1. Develop and refine a CBT-assisted VR prototype for patients with chronic cancer pain (VR-CAN).

Step 2. Conduct a randomized controlled trial to examine the feasibility, acceptability, usability, safety, and initial clinical impact of the developed VR-CAN prototype compared to a tablet-based two-dimensional video control group.

Step 3. Collect and evaluate qualitative post-intervention data on VR-CAN participants' preferences, thoughts, and feelings about the VR-CAN technology and protocol to optimize for a future, larger, fully powered randomized controlled trial.

DETAILED DESCRIPTION:
Over 50% of patients living with cancer experience pain early in the disease course, increasing to at least 75% of patients who have progressed to more advanced stages. Opioid therapies remain a cornerstone to chronic cancer pain management - nevertheless, clinical literature and expert opinion reinforce that maximizing effective, appropriate non-pharmacologic therapies is critical to achieving the best possible pain control, well-being, and return to function. Virtual reality (VR) is a rapidly developing technology that can temporarily immerse individuals in a calm, pleasant environment, and has demonstrated efficacy in acute and chronic pain management settings by providing distraction from pain and lowering pain sensation. Nevertheless, despite growing evidence supporting the efficacy of VR-based interventions for analgesia, few data are available that provide an understanding of its role in mitigating persistent pain in patients with cancer and existing studies have used off-the-shelf VR products that are not evidence-based or designed to meet the unique and complex needs of patients with cancer pain. This collaboration between Duke University and MedStar Health leverages experience conducting clinical trials of VR to mitigate cancer pain in both inpatient and outpatient settings, expertise in the development and implementation of behavioral pain and symptom management interventions for patients with cancer, and experience developing VR applications for healthcare settings. Following the NIH Behavioral Intervention Development Stage Model, the investigators' shared goal is to develop (i.e., patient focus groups, provider and expert interviews, patient beta testing) and pilot test a new VR therapy that integrates evidence-based strategies and is uniquely co-designed by patients living with chronic cancer pain.

Aim 1. Iteratively develop and refine a CBT-assisted VR prototype for patients with chronic cancer pain (VR-CAN) based on literature and the investigative team's research and clinical expertise, and feedback collected via focus groups with patients living with moderate-severe chronic cancer pain and interviews with clinical providers, and experts in the field. Leveraging human factors science, this prototype will then be tested for usability in the lab by patient participants, iteratively modified based on feedback, and then at home by unique participants daily for one week.

Aim 2. Conduct a randomized controlled trial to examine the feasibility, acceptability, usability, safety, and initial clinical impact of the developed VR-CAN prototype compared to a tablet-based two-dimensional video control group.

Aim 3 (Exploratory). Collect and evaluate qualitative post-intervention data on VR-CAN participants' preferences, thoughts, and feelings about the VR-CAN protocol to optimize the VR-CAN protocol that can be efficacy tested in a larger, fully powered randomized controlled trial.

Ultimately, this work has significant potential to decrease burden for a cancer population that experiences high symptom burden and disability.

ELIGIBILITY:
Inclusion Criteria:

* age at least 18 years old
* cancer diagnosis, undergoing treatment
* chronic cancer pain (i.e., cancer pain at least 3 months duration) with baseline pain severity at least 4/10 (where 0=no pain, 10=worst pain)

Exclusion Criteria:

* intractable nausea/vomiting, motion sickness, seizures/epilepsy, and/or cranial structures/abnormalities preventing VR headset use
* moderate-severe pain of non-cancer etiology
* enrolled in another pain study
* unable to complete survey measures or interviews in English or Spanish

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility of device use as assigned | From enrollment to study completion (14 days)
  Protocol adherence (completion of assigned intervention).

SECONDARY OUTCOMES:
Acceptability | From enrollment to study completion (14 days)
  Client Satisfaction Questionnaire (CSQ)
Usability | From enrollment to study completion (14 days)
  System Usability Scale (SUS)
Safety of intervention | From enrollment to study completion (14 days)
  Participants' self-report of side effects
Pain interference | From enrollment to study completion (14 days)
  Pain interference-Short Form (SF)
Profile of Mood States Short Form | From enrollment to study completion (14 days)
  Measures participant psychological distress
Coping Strategies Questionnaire's Pain Catastrophizing subscale | From enrollment to study completion (14 days)
  Measures participant catastrophizing of pain experience
Chronic Pain Self-Efficacy Scale | From enrollment to study completion (14 days)
  Measures participant self-efficacy in pain management
Pain severity | Daily with each use of assigned intervention (during each day of 14 day participation)
  Measures severity of self-reported pain

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - MedStar Health Research Institute, Washington D.C., District of Columbia
  - Duke University School of Medicine, Durham, North Carolina

IPD SHARING:
Plan to Share IPD: Yes
Public use and restricted access study data and associated documentation will be made available to the research community free of charge through the Data Sharing for Demographic Research (DSDR).
Supporting Information: Study Protocol, SAP
Time Frame: Data will become available upon completion of the study and dissemination of findings.
Access Criteria: All deidentified study data that are not designated as restricted use will be made available as public use data to the research community via DSDR. Users of the public use data must register with ICPSR and agree to the Terms of Use, which are designed to protect study participants by limiting data use to scientific research and aggregate statistical reporting, prohibiting attempts to identify study participants, and requiring immediate reporting of any disclosure of study participant identity. Data users also agree not to share or redistribute any data downloads.